CLINICAL TRIAL: NCT00752570
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Study of AMG 386 in Combination With FOLFIRI in Subjects With Previously Treated Metastatic Colorectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20070307
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Cancer; Carcinoma; Colon Cancer; Colorectal Cancer; Gastrointestinal Cancer; Metastases; Metastatic Cancer; Metastatic Colorectal Cancer; Oncology; Rectal Cancer
Keywords: Metastatic Colorectal Cancer; colorectal cancer; colon cancer
MeSH Terms: conditions — Neoplasms; Carcinoma; Colonic Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; Neoplasm Metastasis; Rectal Neoplasms | interventions — trebananib; IFL protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 2 (Placebo Comparator): AMG 386 placebo QW, FOLFIRI Q2W
  Interventions: Drug: AMG 386 Placebo; Drug: FOLFIRI
- 1 (Active Comparator): Arm 1 : AMG 386 10 mg/kg QW, FOLFIRI Q2W
  Interventions: Drug: AMG 386; Drug: FOLFIRI

INTERVENTIONS:
Drug: AMG 386 — AMG 386 (10 mg/kg QW) will be administered until subject develops disease progression, clinical progression, unacceptable toxicity, or withdraws consent.
  Arms: 1
Drug: AMG 386 Placebo — AMG 386 placebo QW will be administered until subject develops disease progression, clinical progression, unacceptable toxicity, or withdraws consent.
  Arms: 2
Drug: FOLFIRI — Administration of FOLFIRI chemotherapy will commence on day 1 of each dosing week following the administration of AMG 386.
  FOLFIRI Q2W regimen: irinotecan 180 mg/m2 IV over 90 (+-15) minutes on Day 1, leucovorin 400 mg/m2 IV over 2 hrs on Day 1, 5 FU 400mg/m2 IV bolus, followed by 2400 mg/m2 continuous IV infusion over 46 hrs +- 2 hours.
  FOLFIRI will be administered until disease progression, FOLFIRI intolerability, death, or study withdrawal by the subject, investigator, or sponsor, whichever occurs earliest.

SUMMARY:
This clinical trial will compare the efficacy and safety of the combination of AMG 386 and FOLFIRI with FOLFIRI alone in second line treatment of metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum in patients who are presenting with metastatic disease
* One and only one prior chemotherapy regimen for metastatic disease consisting of the combination of a fluoropyrimidine-based chemotherapy and an oxaliplatin-based chemotherapy. Prior adjuvant chemotherapy used prior to the onset of metastatic disease is permitted
* At least one uni dimensionally measurable lesion per modified RECIST criteria. All sites of disease must be evaluated <= 28 days before randomization
* Radiographically documented disease progression per modified RECIST criteria either while receiving or <= 6 months after the last dose of prior chemotherapy regimen for metastatic disease
* ECOG performance status of 0 or 1
* Man or woman >= 18 years of age
* Adequate end organ assessments by laboratory studies (hematological and chemistries)
* Life expectancy >= 3 months

Exclusion Criteria:

* Exclude subjects with a history of prior malignancy, except:

  * Malignancy treated with curative intent and with no known active disease present for >= 3 years before enrollment and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
* Prior irinotecan therapy
* Systemic chemotherapy, hormonal therapy, or immunotherapy <= 21 days prior to randomization
* Experimental or approved proteins/antibodies (eg, bevacizumab) <= 30 days prior to randomization
* Clinically significant cardiac disease within 12 months prior to randomization, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication, percutaneous transluminal coronary angioplasty/stent
* Known allergy or hypersensitivity to irinotecan, 5 FU (known dihydropyrimidine dehydrogenase deficiency) or leucovorin
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhea (defined as >= CTC grade 2 [CTCAE version 3.0])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To estimate the treatment effect as measured by progression free survival (PFS) in subjects treated with AMG 386 + FOLFIRI relative to subjects treated with FOLFIRI + placebo. | The time frame will be event driven and will occur when 100 subjects have experienced a PFS event (radiographic disease progression or death).

SECONDARY OUTCOMES:
To evaluate other measures of efficacy or clinical response including objective response rate (ORR), duration of response (DOR), overall survival (OS) in subjects treated with AMG 386 + FOLFIRI relative to subjects treated with FOLFIRI + placebo | Treatment phase or until disease progression
To evaluate progression free survival and measures of efficacy by KRAS status | Treatment phase
To evaluate patient reported outcomes (PROs), relative dose intensity, incidence of anti AMG 386 antibody formation, pharmacokinetics of AMG 386 (Cmax and AUC) and safety (incidence of AEs and significant laboratory changes) | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Peeters M, Strickland AH, Lichinitser M, Suresh AV, Manikhas G, Shapiro J, Rogowski W, Huang X, Wu B, Warner D, Jain R, Tebbutt NC. A randomised, double-blind, placebo-controlled phase 2 study of trebananib (AMG 386) in combination with FOLFIRI in patients with previously treated metastatic colorectal carcinoma. Br J Cancer. 2013 Feb 19;108(3):503-11. doi: 10.1038/bjc.2012.594. Epub 2013 Jan 29. PMID 23361051
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com